CLINICAL TRIAL: NCT06063655
Title: A Randomized, Placebo Controlled, Semi-Blind, Crossover Study to Evaluate the Effects of Two Novel Hydration Beverage Formulas on Rehydration in Adults
Brief Title: Effects of Two Novel Hydration Beverage Formulas on Rehydration in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2023-416
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: A Randomized, Placebo Controlled, Semi-Blind, Crossover Study
Who Masked: Participant
Masking Description: Subjects will be assigned conditions via a code (A, B, C)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Water, Hydration Multiplier, Sugar-Free (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: water, Liquid IV Hydration Multiplier, and Liquid IV Sugar-Free Hydration Multiplier.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier
- Water, Sugar-Free, Hydration Multiplier (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: water, Liquid IV Sugar-Free Hydration Multiplier, and Liquid IV Hydration Multiplier.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier
- Hydration Multiplier, Sugar-Free, Water (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: Liquid IV Hydration Multiplier, Liquid IV Sugar-Free Hydration Multiplier, and water.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier
- Hydration Multiplier, Water, Sugar-Free (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: Liquid IV Hydration Multiplier, water, and Liquid IV Sugar-Free Hydration Multiplier.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier
- Sugar-Free, Water, Hydration Multiplier (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: Liquid IV Sugar-Free Hydration Multiplier, water, and Liquid IV Hydration Multiplier.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier
- Sugar-Free, Hydration Multiplier, Water (Experimental): Subjects will undergo three 90-min cycling bouts at 70-80% maximal hear rate, 86-89 degrees Fahrenheit, and approximately 50% relative humidity spaced 1-2 weeks apart. Subjects will be provided with a different test drink after each cycling bout at an amount equivalent to150% of sweat losses and evaluated for rehydration.
  Subjects randomly assigned to this arm will be provided with the experimental/placebo conditions in the following order: Liquid IV Sugar-Free Hydration Multiplier, Liquid IV Hydration Multiplier, and water.
  Interventions: Dietary Supplement: Control: Water; Dietary Supplement: Liquid IV hydration multiplier; Dietary Supplement: Liquid IV sugar-free hydration multiplier

INTERVENTIONS:
Dietary Supplement: Control: Water — Water will be provided to subject divided into 3 equal portions with each portion consumed over 10 minutes with 15 minutes between portions (rehydration period of 1 hour).
Dietary Supplement: Liquid IV hydration multiplier — Liquid IV hydration multiplier will be provided to subject divided into 3 equal portions with each portion consumed over 10 minutes with 15 minutes between portions (rehydration period of 1 hour).
Dietary Supplement: Liquid IV sugar-free hydration multiplier — Liquid IV sugar-free hydration multiplier will be provided to subject divided into 3 equal portions with each portion consumed over 10 minutes with 15 minutes between portions (rehydration period of 1 hour).

SUMMARY:
The electrolyte test products are composed of powder and provided in individual stick packs with 5 vitamins including Vitamins B3, B5, B6, B12 and Vitamin C. The products are gluten-, soy-, and dairy-free, and provide electrolytes at concentrations well below the daily value (DV). The DV tells us how much a particular nutrient in a serving of a food product contributes to a daily diet, based on a standard 2000 calorie diet. Despite what the name suggests, this product is taken orally, not intravenously. These packets contain a small percentage of the needed total daily electrolytes but adequate amounts to replace lost electrolytes as a result of physical activity.

The products will be consumed following a 90-minute bout of cycling exercise at a moderate intensity of 70-80% max heart rate, at 30-32°C (86-89°F) and 50 ± 5% relative humidity. This same exercise duration and room temperature has been used in a recent study, which also utilized the same body temperature monitoring device as proposed in the present study. The purpose of the exercise bout is to simulate what many individuals are exposed to when exercising in the heat and to moderately dehydrate subjects, as would be the case during a moderate run or cycling event in exercise-trained individuals.

Subjects will report to the lab on three separate occasions to consume one of the 3 drinks (hydration multiplier, sugar-free hydration matrix, or water), in random order. The drinks will be consumed during the post-exercise period (30 minutes following the completion of exercise).

DETAILED DESCRIPTION:
Maintaining adequate hydration is essential to optimal health, as well as athletic performance. When individuals exercise (in particular in a warm environment), they can lose excessive amounts of fluids along with necessary electrolytes (e.g., sodium, potassium, chloride) through sweating. With dehydration, individuals may feel sluggish and can experience impaired physical performance.

The use of electrolytes (sodium in particular) has been used for decades to aid athlete hydration and has led to the development of various sport drinks (e.g., Gatorade, Powerade) -which also include small amounts of carbohydrate.

This study will evaluate the hydration effects of two electrolyte products dissolved in water (Hydration Multiplier and Sugar-Free Hydration Multiplier) compared to a placebo (water). The nutrient composition of the Sugar-Free hydration Multiplier is similar to the Liquid IV Hydration Multiplier product currently on the market but without sugar content.

The electrolyte test products are composed of powder and provided in individual stick packs with 5 vitamins including Vitamins B3, B5, B6, B12 and Vitamin C. The products are gluten-, soy-, and dairy-free, and provide electrolytes at concentrations well below the daily value (DV). The DV tells us how much a particular nutrient in a serving of a food product contributes to a daily diet, based on a standard 2000 calorie diet. Despite what the name suggests, this product is taken orally, not intravenously. These packets contain a small percentage of the needed total daily electrolytes but adequate amounts to replace lost electrolytes as a result of physical activity.

The products will be consumed following a 90-minute bout of cycling exercise at a moderate intensity of 70-80% max heart rate, at 30-32°C (86-89°F) and 50 ± 5% relative humidity. This same exercise duration and room temperature has been used in a recent study, which also utilized the same body temperature monitoring device as proposed in the present study. The purpose of the exercise bout is to simulate what many individuals are exposed to when exercising in the heat and to moderately dehydrate subjects, as would be the case during a moderate run or cycling event in exercise-trained individuals.

Subjects will report to the lab on three separate occasions to consume one of the 3 drinks (hydration multiplier, sugar-free hydration matrix, or water), in random order. The drinks will be consumed during the post-exercise period (30 minutes following the completion of exercise).

This study design and outcomes have been similarly used in previous rehydration studies that utilized exercise in heat to induce ~2% body weight loss with different test products . This study will help further the knowledge on how different formulations of hydration beverages (e.g., different carbohydrate and electrolyte compositions) alter rehydration following exercise. It is hypothesized that both test products will provide improved rehydration above water alone during the post-exercise period. Moreover, it is believed that the sugar free product may improve hydration similar to the standard Hydration Multiplier.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 17.0-29.9 kg/m2 (not obese)
* Resting heart rate less than 90 beats per minute; although, if less than 40 beats per minute subject must get clearance from a medical professional
* Not hypertensive (Systolic <140 mmHg and Diastolic <90 mmHg)
* Have not had in the 3 months prior to screening or planning to have a major surgery during study period
* Physically capable and willing to ingest the assigned amount of fluid while cycling and at rest for visits 3, 4, and 5
* Must be moderately trained; engage in moderate intensity, intermittent, or steady-state exercise at least 3 days per week for at least one hour at a time.
* Willing to maintain the same level of physical activity throughout the study period, except during the 24 hour period prior to each study visit.
* Achieve a peak maximal oxygen consumption at screening that is at least 60% of their age and gender matched normative value per American College of Sports Medicine recommendations.
* Capable of completing 90 minutes of self-paced stationary cycling (~70-80% max heart rate) in a heated environmental chamber (~30-32°C (86-89°F) with ~50% RH).
* Can drink a minimum of 2.0 L fluid (if female) or 2.5 L fluid (if male) the day prior to test visits
* For visits 3-5, subjects must have a urine specific gravity less than 1.020.
* For visit 3-5, subject must not have exercised within 24 hours of visit
* Consume no more than two standard alcoholic drinks per day on a regular basis and during study period.
* Maintain diet, exercise, BMI, medication, and dietary supplements throughout study period as changes may alter hydration and electrolyte levels and result in changes to outcome measures.

Exclusion Criteria:

* If female, lactating, pregnant or planning to become pregnant during the study.
* Have a known sensitivity or allergy to any of the study products
* Have a history of diabetes
* Have a history of known cardiovascular disease
* Have a history of a diagnosis of celiac disease, chronic pancreatitis, steatorrhea, unstable thyroid disease, immune disorder (i.e., HIV/AIDS), cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
* Have an active or uncontrolled diseases or conditions
* Have had a current or previous Corona virus disease 2019 diagnosis in the three months prior to screening.
* Have any medical conditions that may impact ability to exercise or ability to ingest prescribed fluid volume as determined by the study nurse, including infection or illness
* Weighing less than 80 lbs at any visit; although very unlikely, we need to maintain this cut off, as too low a body mass is unhealthy.
* Has taken within 30 days or within seven half-lives (whichever is longer) of first test visit: selective serotonin uptake inhibitors (SSRI), Apremilast, caffeine-containing drugs, Corticosteroids (systemic use), Decongestants, Diuretics, Laxatives, Muscle relaxants, Opioid painkillers, Statins, Oral antibiotics
* Has taken within 30 days of first test visit: Calcium, Dandelion, Lithium orotate, Potassium citrate, Watercress, Inhalables smokables, or the like cigarettes, vaporizers, water pipes, or cannabis
* Has taken within 24 hours prior to test visit: Alcohol, Caffeine (including coffee, tea, energy drinks, etc. prohibited in the 12hrs prior to each dose of the study product), Laxatives, Diuretics, or Sports drinks (electrolyte drinks)
* received or use test product(s) in another research study in the 28 days prior to baseline visit (Familiarization, Visit/Visit 2), or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of the current study.
* have any other active or unstable medical conditions or use medications, supplements, or therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | baseline (prior to cycling)
  body weight will be measured using a digital scale
Body weight | 0 minutes after 90-minute cycle bout
  body weight will be measured using a digital scale
Body weight | 30 minutes after cycling
  body weight will be measured using a digital scale
Body weight | 4 hours and 30 minutes after cycling
  body weight will be measured using a digital scale
Urine Volume | baseline (prior to cycling)
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 0 minutes after cycling
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 30 minutes after cycling
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 1 hour 30 minutes after cycling (following rehydration period)
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 2 hours 30 minutes after cycling
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 3 hours 30 minutes after cycling
  urine will be collected in a tray and then weighed on a digital scale
Urine Volume | 4 hours 30 minutes after cycling
  urine will be collected in a tray and then weighed on a digital scale
Urine osmolality | baseline (prior to cycling)
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 0 minutes after cycling
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 30 minutes after cycling
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 1 hour 30 minutes after cycling (following rehydration period)
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 2 hour 30 minutes after cycling (following rehydration period)
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 3 hour 30 minutes after cycling (following rehydration period)
  Osmolality will be determined from a urine sample collected in a tray
Urine osmolality | 4 hour 30 minutes after cycling (following rehydration period)
  Osmolality will be determined from a urine sample collected in a tray
Urine specific gravity | first morning urine (~2 hours before visit)
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | baseline (before cycling)
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 0 minutes after cycling
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 30 minutes after cycling
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 1 hour 30 minutes after cycling (following rehydration period)
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 2 hour 30 minutes after cycling (following rehydration period)
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 3 hour 30 minutes after cycling (following rehydration period)
  specific gravity will be determined using a refractometer from a urine sample collected
Urine specific gravity | 4 hour 30 minutes after cycling (following rehydration period)
  specific gravity will be determined using a refractometer from a urine sample collected
Plasma Osmolality | baseline (before cycling)
  Blood will be collected to determine plasma osmolality
Electrolyte levels | baseline (before cycling)
  electrolyte levels will be measured in blood
Percent plasma volume | baseline (before cycling)
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 30 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 30 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 30 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 60 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 60 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 60 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 120 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 120 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 120 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 150 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 150 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 150 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 210 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 210 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 210 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.
Plasma Osmolality | 270 minutes post cycling
  Blood will be collected to determine plasma osmolality
Electrolyte levels | 270 minutes post cycling
  electrolyte levels (Sodium, potassium, chloride, and carbon dioxide total) will be measured in blood (millimoles per liter)
Percent plasma volume | 270 minutes post cycling
  Percent plasma volume will be determined by measuring hematocrit and hemoglobin in blood.

SECONDARY OUTCOMES:
Body temperature | Every 10 minutes during cycling
  Body temperature will be monitored during cycling
Heart rate | Every 10 minutes during cycling
  Heart rate will be monitored during cycling
Rate of Perceived Exertion | Every 10 minutes during cycling
  Rate of Perceived Exertion using a Borg scale from 6 (easy) to 20 (maximal effort) will be reported during cycling
maximal oxygen consumption | At screening
  maximal oxygen consumption will be determined via a cycling test
Height | At screening
  Height will be measured using a stadiometer
Weight | At screening
  Weight will be determined using a digital scale
Waist/Hip ratio | At screening
  Waist/Hip ratio will be determined by measuring each circumference with a tape measure
Resting Diastolic Blood Pressure | At screening
  Diastolic blood pressure will be measured after a 10 minute rest sitting using a digital machine
Resting Systolic Blood Pressure | At screening
  Systolic blood pressure will be measured after a 10 minute rest sitting using a digital machine
Heart Rate | At screening
  Heart Rate will be measured after a 10 minute rest sitting using a digital machine

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States